CLINICAL TRIAL: NCT03615456
Title: Sutureless Thyroidectomy Versus Conventional Thyroidectomy: Prospective Randomized Clinical Trial
Brief Title: Sutureless Versus Conventional Thyroidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Sameh Emile, Assistant professor of surgery, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: mansoura62
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Goiter
MeSH Terms: conditions — Goiter

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional thyroidectomy (Active Comparator): Thyroidectomy with ligation and division of thyroid vessels
  Interventions: Procedure: Conventional thyroidectomy
- Harmonic scalpel thyroidectomy (Active Comparator): Thyroidectomy with sealing of thyroid vessels using harmonic scalpel
  Interventions: Procedure: Harmonic scalpel thyroidectomy

INTERVENTIONS:
Procedure: Conventional thyroidectomy — Thyroid vessels are ligated with sutures and divided
  Arms: Conventional thyroidectomy
Procedure: Harmonic scalpel thyroidectomy — Thyroid vessels are sealed using harmonic scalpel device
  Arms: Harmonic scalpel thyroidectomy

SUMMARY:
This study was prospective randomized double-blinded clinical trial on patients with thyroid disease who underwent thyroidectomy in the general surgery department, Mansoura university hospitals during the period of February 2017 to February 2018.Two techniques for vascular sealing were compared: conventional tying and harmonic scalpel

ELIGIBILITY:
Inclusion Criteria:

Patients of both genders aging above 18 years presented with primary thyroid diseases requiring thyroidectomy including:

* Solitary thyroid nodule (STN)
* Multinodular goiter
* Controlled toxic goiter
* Inflammatory goiter (thyroiditis)
* Early-stage thyroid cancer.

Exclusion Criteria:

* Patients unfit for surgery
* patients unwilling to participate in the study
* Pregnant women
* Thyroid cancer with lymph node or distant metastasis.
* Patients with psychiatric disturbances.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-05-12 (Actual)

PRIMARY OUTCOMES:
Volume of postoperative drainage | At 24 hours after surgery
  The volume of fluid drained in the suction drain placed in the neck in milliliters

CONTACTS AND LOCATIONS:
Overall Officials: Sabry Mahmoud, M.D., Study Chair — Mansoura University
Locations (1):
- Mansoura university hospital, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No